CLINICAL TRIAL: NCT02333721
Title: Study on Long-term Outcome of Laparoscopic Spleen-Preserving D2 Lymphadenectomy With and Without No. 10 Lymph Node Dissection for Advanced Gastric Cancer
Brief Title: Study on Laparoscopic Spleen-Preserving No. 10 Lymph Node Dissection for Advanced Middle or Upper Third Gastric Cancer
Acronym: LSPLN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director, Principal Investigator, Clinical Professor, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-002
Record Dates: First submitted 2014-12-25; First posted 2015-01-07 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Laparoscopy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D2 Lymphadenectomy including No. 10 (Experimental): Laparoscopic total gastrectomy with D2 lymphadenectomy including spleen-preserving No. 10 lymph node dissection will be performed for the treatment of patients assigned to this group
  Interventions: Procedure: D2 lymphadenectomy including No. 10
- D2 lymphadenectomy excluding No. 10 (Active Comparator): Laparoscopic total gastrectomy with D2 lymphadenectomy excluding spleen-preserving No. 10 lymph node dissection will be performed for the treatment of patients assigned to this group
  Interventions: Procedure: D2 lymphadenectomy excluding No. 10

INTERVENTIONS:
Procedure: D2 lymphadenectomy including No. 10 — After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, Laparoscopic total gastrectomy with D2 lymphadenectomy including spleen-Preserving No. 10 Lymph Node Dissection will be performed with curative treated intent. The type of reconstruction will be selected according to the surgeon's experience and anastomotic procedure is performed extracorporeally using a mini-laparotomy
  Arms: D2 Lymphadenectomy including No. 10
Procedure: D2 lymphadenectomy excluding No. 10 — After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, Laparoscopic total gastrectomy with D2 lymphadenectomy excluding spleen-Preserving No. 10 Lymph Node Dissection will be performed with curative treated intent. The type of reconstruction will be selected according to the surgeon's experience and anastomotic procedure is performed extracorporeally using a mini-laparotomy
  Arms: D2 lymphadenectomy excluding No. 10

SUMMARY:
The purpose of this study is to explore the short-term, long-term and oncological outcomes of laparoscopic spleen-preserving No. 10 lymph node dissection in a left-sided approach for advanced middle or upper third gastric cancer not invading greater curvature.

DETAILED DESCRIPTION:
A prospective randomized comparison of laparoscopic spleen-preserving No. 10 lymph node dissection for gastric cancer will be performed, to evaluate the short-term, long-term and oncological outcomes. The evaluation parameters are perioperative clinical efficacy, postoperative life quality, immune function and 3-year survival and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years
* Primary proximal gastric adenocarcinoma not invading greater curvature (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
* cT2-4a, N0-3, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition
* No distant metastasis is observed. And the spleen, pancreas or other adjacent organs are not involved by the tumor.
* Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
* American Society of Anesthesiology score (ASA) class I, II, or III
* Written informed consent

Exclusion Criteria:

* Women during pregnancy or breast-feeding
* Severe mental disorder
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
* Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging
* History of other malignant disease within past five years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within past six months
* History of cerebrovascular accident within past six months
* History of continuous systematic administration of corticosteroids within one month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of predicted values

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 536 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months

SECONDARY OUTCOMES:
Morbidity and mortality | 30 days; 36 months
  The early postoperative complication and mortality are defined as the event observed within 30 days after surgery, while the time frame for late complication is the period from postoperative day 31th to the end of month 36th.
3-year overall survival rate | 36 months
  3-year overall survival rate
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type
Time to first ambulation | 10 days
  The data of postoperative recovery course.
Rates of splenectomy | 1 day
  splenectomy performing by severe injury to the splenic vessels
Rates of injury to splenic vessels | 1 day
  intraoperative injury to the splenic vessels
The number of lymph node dissection | 1 day
  The total number of lymph node dissection and the number of lymph node dissection in each station
The variation of weight | 12 months
  The variation of weight on postoperative 3, 6, 9 and 12 months
The daily highest body temperature | 7 days
  The daily highest body temperature before discharge
Time to first flatus | 10 days
  The time to first flatus
Time to first liquid diet | 10 days
  The time to first liquid diet
Time to soft diet | 10 days
  The time to soft diet
Duration of hospital stay | 10 days
  Duration of hospital stay
The amount of abdominal drainage | 10 days
  The amount of abdominal drainage
Blood transfusion | 10 days
  Perioperative blood transfusion
The number of positive lymph nodes | 1 day
  The number of positive lymph nodes
Intraoperative lymph node dissection time | 1 day
  intraoperative No.10 lymph node dissection time includes infrapyloric area lymph node,suprapancreatic area lymph node,splenic hilar area lymph node, cardial area lymph node)
Intraoperative blood loss | 1 day
  Intraoperative blood loss
Intraoperative injury | 1 day
  Intraoperative injury
The amount of use of titanium clip | 1 day
  The amount of use of titanium clip
The rate of conversion to laparotomy | 1 day
  The rate of conversion to laparotomy
The variation of cholesterol | 12 months
  The variation of cholesterol on postoperative 3, 6, 9 and 12 months
The variation of albumin | 12 months
  The variation of albumin on postoperative 3, 6, 9 and 12 months
The results of endoscopy | 12 months
  the results of endoscopy on postoperative 3 and 12 months
The values of white blood cell count | 7 days
  the values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
The values of hemoglobin | 7 days
  and the values of hemoglobin from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
The values of C-reactive protein | 7 days
  and the values of C-reactive protein from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
The values of prealbumin | 7 days
  and the values of prealbumin from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
The values of relevant immune cytokines | 7 days
  and the values of relevant immune cytokines including T cell percentage, T-helper lymphocytes (CD4+) percentage, T-suppressor lymphocytes (CD8+) percentage, natural killer (NK) cells percentage from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
The Surgery Task Load Index (SURG-TLX) | 1 days
  Surgeons were required to complete one modified SURG-TLX questionnaire for each procedure.
Lymph node noncompliance rate | 1 days
  Lymph node noncompliance was defined as the absence of lymph nodes that should have been excised from more than 1 lymph node station. Major lymph node noncompliance was defined as more than 2 intended lymph node stations that were not removed.
Technical performance | 1 days
  Technical performance were assessed by the Objective Structured Assessments of Technical Skills (OSATS) and the Generic Error Rating Tool.

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, M.D.,Ph.D., Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhong Q, Zhang ZQ, Yan YQ, Li YF, He QC, Zheng CH, Chen QY, Huang CM. [Long-term oncological safety of robotic total gastrectomy for locally advanced proximal gastric cancer: a 5-year noninferiority comparison based on the FUGES-014 study]. Zhonghua Wei Chang Wai Ke Za Zhi. 2025 Aug 25;28(8):886-894. doi: 10.3760/cma.j.cn441530-20250610-00218. Chinese. PMID 40850834
- [Derived] Xu BB, Zheng HL, Chen CS, Xu LL, Xue Z, Wei LH, Zheng HH, Shen LL, Zheng CH, Li P, Xie JW, Lin JX, Zheng YH, Huang CM. Development and validation of a preoperative radiomics-based nomogram to identify patients who can benefit from splenic hilar lymphadenectomy: a pooled analysis of three prospective trials. Int J Surg. 2024 Jul 1;110(7):4053-4061. doi: 10.1097/JS9.0000000000001337. PMID 38980664
- [Derived] Lin JX, Xu BB, Zheng HL, Li P, Xie JW, Wang JB, Lu J, Chen QY, Cao LL, Lin M, Tu RH, Huang ZN, Lin JL, Yao ZH, Zheng CH, Huang CM. Laparoscopic Spleen-Preserving Hilar Lymphadenectomy for Advanced Proximal Gastric Cancer Without Greater Curvature Invasion: Five-Year Outcomes From the Fuges-02 Randomized Clinical Trial. JAMA Surg. 2024 Jul 1;159(7):747-755. doi: 10.1001/jamasurg.2024.1023. PMID 38691353
- [Derived] Lin JX, Lin JP, Wang ZK, Li P, Xie JW, Wang JB, Lu J, Chen QY, Cao LL, Lin M, Tu RH, Lin GT, Huang ZN, Lin JL, Zheng HL, Lin GS, Huang CM, Zheng CH. Assessment of Laparoscopic Spleen-Preserving Hilar Lymphadenectomy for Advanced Proximal Gastric Cancer Without Invasion Into the Greater Curvature: A Randomized Clinical Trial. JAMA Surg. 2023 Jan 1;158(1):10-18. doi: 10.1001/jamasurg.2022.5307. PMID 36383362